CLINICAL TRIAL: NCT07092072
Title: One-year Efficacy and Tolerance of Myofix Spectacles for the Control of Myopia Progression
Brief Title: Efficacy and Tolerance of Full Field Peripheral Defocus Spectacles for the Control of Myopia Progression (Myofix Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novar Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Registration No. 8638/23; Registration No. 8638 (Other: Ethics Committee of the Argentine Society of Ophthalmology)
Record Dates: First submitted 2025-07-18; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myopia Progression
Keywords: Myopia control spectacles, full field defocus design

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MYOPIA TREATED (Experimental): MYOPIC CHILDREN TREATED WITH MYOFIX SPECTACLES
  Interventions: Device: MYOFIX FULL FIELD PERIPHERAL DEFOCUS SPECTACLE

INTERVENTIONS:
Device: MYOFIX FULL FIELD PERIPHERAL DEFOCUS SPECTACLE — This is a plus peripheral add spectacle with the central part for the myopic correction.

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the use of a new model of spectacles designed to control the progression of myopia in childhood. School myopia in children is mainly produced by increased ocular growth. This new spectacle design is based in the fact that positive lenses in front of eyes produce changes that decrease ocular growth. It consists of a full field peripheral positive defocus lens and a central section for the distance correction. The study is designed to evaluate tolerance and efficacy of this new lens in myopic children along a two year period.

DETAILED DESCRIPTION:
The Myofix Defocus Study is a longitudinal, prospective, interventional, non-randomized research study intended to evaluate the tolerability and effectiveness of the use of spectacles with special design to control the progression of myopia during childhood. This field study included children aged 8 to 15 years old who voluntarily agreed to use the Defocus Spectacles for one year. A pair of spectacles (Myofix, Novar, Argentina) with frames (Usual, Argentina) were provided free of charge to all children studied for one year with the special addendum of peripheral defocus treatment. Children are instructed to wear the glasses the whole day every day of the week including Saturdays and Sundays.The Argentinian Defocus Spectacle lens design preserves the principle of the original design presented by Carly Lam et al., which consisted of a 9 mm central zone for distance correction and a +3.50 diopters defocus correction ring of lenslets laying between 9 and 32 mm diameter to act primarily on the para foveal zone that detects the defocus that governs the growth of the eye. Instead of micro peripheral defocus lenses in the 32 mm diameter ring zone with treatment, our model has a uniform peripheral +/+3.50 diopters power zone add. As it is known that 30-40 minutes of exposure to myopic defocus modifies the axial length (measured with Lenstar) by approximately 10-15 microns due to changes in choroidal thickness, the national design has been tested on 17 volunteer subjects showing a significant change of 11 microns shortening in the axial length of their eyes, such that that pilot study suggested the lenses could be effective in arresting the progression of myopia, as changes in the choroid are the first events in the retinal message that manages ocular growth. For comparing the outcomes of this study two virtual control groups in American children will be considered. One control group will be taken from a study in US giving children diluted atropine drops for myopia control. The placebo treated arm of this group will be considered. The other control group will be a cohort of children followed up in Argentina with cycloplegic refractions one year before the pandemic closeup began.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 16 years who voluntarily agreed to use the Defocus spectacles for one year.
* A consecutive series of children diagnosed with myopia, attending accredited private practice ophthalmology clinics across Argentina.
* Absence of ocular pathology other than myopia,
* Spherical equivalent (SE = sphere + [cylinder/2]) between ≤-0.50 D and -5.00 D
* Astigmatism less than -2.00 D
* Anisometropia less than -1.00 D
* Keratometry less than 47.00 D in the steepest meridian
* The corrected distance visual acuity based on subjective refraction was required to be 0.1 logMAR (20/25 Feet Snellen) or better in each eye.

Exclusion Criteria:

* Myopia with onset before the age of 6 years,
* Any genetic syndromes,
* Current medical treatment for myopia other than single vision spectacle correction.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
RATE OF MYOPIA PROGRESSION IN DIOPTERS | 12 MONTHS AND 24 MONTHS FOLLOW UP PLANNED
  THE AMOUNT OF DIOPTERS OF MYOPIC PROGRESSION IN ONE YEAR FOLLOW UP MEASURED WITH CYCLOPLEGIC REFRACTIONS

CONTACTS AND LOCATIONS:
Locations (1):
- Drs. Iribarren Eye Consultants, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
There are plans to share individual participant data if any investigator in the area of myopia control research asks us about the data.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD and supporting information will be available after the study is finished and published with no time limit.
Access Criteria: Any researcher in myopia control area may ask for the data. The data will be provided in an SSPS dataset, send at their formal request.

REFERENCES:
- [Background] De Tomas M, Kotlik C, Szeps A, Impagliazzo R, Iribarren R. New Spectacles for Myopia Control. Oftalmol Clin Exp. 2022; 15: 240-7.
- [Background] Iribarren R SA, Kotlik C, Laurencio L, De Tomas M, Impagliazzo R, Martin G. Short-Term Axial Length Changes in Myopic Eyes Induced by Defocus Spectacles for Myopia Control. Photonics 2023; 10: 668.
- [Background] De Tomás M SA, Martín G, Saracco G, Lanca C, Iribarren R. Effect of vertex distance in the treatment area of myopia control spectacles. Oftalmol Clin Exp 2024; 17: e547-e53.
- [Background] Saracco G AM, De Tomás M, Martín G, Iribarren R. Development of a frame adaptation for myopia control spectacles. Oftalmol Clin Exp 2025; 18: e195-e201.
- [Result] Szeps A KC, Fernández Irigaray L, Saracco G, De Tomas M, Martin G, Iribarren R. Baseline data in the study on the tolerance and efficacy of peripheral defocus spectacles for the control of myopia progression in Argentina (Myofix Defocus Study). Oftalmol Clin Exp 2024; 17: 352-8.
- [Derived] Iribarren R, Szeps A, Kotlik C, de Tomas M, Martin G, Rozema J, Lanca C. One-Year Efficacy and Tolerance of Myofix Defocus Spectacles for Control of Myopia Progression. Ophthalmol Ther. 2025 Nov 12. doi: 10.1007/s40123-025-01270-4. Online ahead of print. PMID 41222872

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-03-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT07092072/Prot_SAP_ICF_000.pdf